CLINICAL TRIAL: NCT02740049
Title: In Vitro Evaluation of a Novel Drug on Airway Epithelial Cells Obtained From Participants With Severe Asthma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Vectura Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15IC2844
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: Epithelial Cells
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Astma patients (Experimental): Participant undergoes a bronchoscopy to isolate epithelial cells
  Interventions: Drug: VR588

INTERVENTIONS:
Drug: VR588 — Evaluation of the efficacy of a novel JAK/STAT inhibitor, VR588, in isolated epithelial cells from asthma patients

SUMMARY:
Asthma is a long term disease of the lungs. In asthma patients the sensitive airway tubes narrow in reaction to something that irritates the airways such as allergens or environmental pollutants. There is currently no cure for asthma and new medicines or combinations of medicines are needed that will be of benefit to patients particularly those with a more severe disease.

Activation of certain signal molecules inside the lung cells may participate in the development of asthma and the response to allergens. Blocking these signal molecules specifically with medicines might therefore be beneficial in the treatment of asthma. In this study we want to test a new medicine that specifically targets a subset of signal molecules that are associated with the allergen response in the lung. In particular, we want to test this medicine on cells obtained from the lungs of asthma patients. Understanding the effects of this new medicine on these asthmatic lung cells will give vital information on how this new medicine works before we can test it in asthma patients.

DETAILED DESCRIPTION:
Asthma and COPD are chronic inflammatory diseases of the airway although the precise cells and mediators involved are distinct. Both diseases are characterised by airway hyperresponsiveness (AHR) in response to exogenous stimuli such as allergens in asthma or environmental pollutants. There is currently no cure for asthma and new drugs or combinations of drugs are needed that will be of benefit to patients particularly those with more severe disease.

Activation of JAK/STAT pathways may participate in the pathogenesis of asthma. STAT1 and STAT6 expression is elevated in animal models of asthma and in the lower airways of some but not all patients. STAT6 is activated by key cytokines involved in asthma such as IL-13 in primary human bronchial epithelial cells. In addition, baseline phospho-STAT1 and phospho-STAT6 levels are increased in systemic T cells from steroid naïve asthmatics and the Th2 cytokines IL-4, IL-13 and TSLP activate STAT1 and STAT6 in a number of airway cells. In animal models of allergen-induced AHR, airway inflammation including CXCL9 and CXCL10 involves STAT1. In addition, STAT6 knockout mice have no response to IL-4, do not develop Th2 cells in response to IL-4, and fail to produce IgE, bronchial hyperresponsiveness or BAL eosinophilia after allergen sensitization. The expression of CCL11, CCL17 and CCL22 also involves STAT6 in these models.

Importantly, STAT1 is a critical signalling molecule involved in the production of type I IFNs (α/β), IFN-γ and for resistance to viral respiratory infections. JAK/STATs inhibitors have proved effective in clinical trials for rheumatoid arthritis and inflammatory bowel disease.

Therefore, we propose to use the primary airway epithelial cell culture model grown at air:liquid interface (ALI culture) to evaluate the efficacy of a novel JAK/STAT inhibitor, VR588, against CP-690550 and fluticasone proprionate (FP) in suppressing inflammatory readouts induced by IL-13 and by TNF/IFN.

ELIGIBILITY:
Inclusion Criteria:

All patients must be able to give informed consent.

The definition of severe asthma will be on the basis of:

1. Treatment: High dose of ICS ± OCS ≥ 1000mcg FP daily or equivalent plus one other controller medication.
2. Disease Control: Uncontrolled (GINA guidelines), three or more of the following present in any week in the preceding 4 weeks:

   1. Daytime symptoms more than twice per week
   2. Any limitation of activities
   3. Nocturnal symptoms once or more per week
   4. Need for reliever treatment more than twice per week
   5. Prebronchodilator FEV1 <80% predicted or personal best AND/OR Frequent severe exacerbations (≥2 per year requiring high dose OCS or doubling of maintenance dose for at least three days or requiring hospitalisation).
3. Asthma Diagnosis:

Improvement in FEV1 ≥ 12% or 200ml predicted after inhalation of 400mcg salbutamol OR Diurnal variation in PEF: amplitude % mean of twice daily PEF > 8% OR Decrease in FEV1 ≥ 12% and >200ml within 4 weeks after tapering treatment with one or more of the following drugs: ICS, OCS, LABA, SABA PLUS A history of wheeze occurring spontaneously or on exertion.

Exclusion Criteria:

1. Patients with a FEV1 < 1L
2. Any other active lung condition
3. Subjects unable to give consent

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fan Chung, MD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant diagnosed with severe asthma were recruited from clinics at the Royal Brompton hospital between January 2016 and September 2016.
Period: Overall Study
Arm/Group | Astma Patients
Started | 9
Completed | 8
Not Completed | 1
Not completed — Isolated cells did not grow sufficiently | 1

BASELINE CHARACTERISTICS:
Arm/Group | Astma Patients
Number analyzed (Participants) | 9
Age, Customized [Mean (Standard Deviation); unit: years]
  Participants | 51.9 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian | 1
  White | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9

OUTCOME MEASURES:

1. Primary Outcome: Concentration (pg/ml) of CXCL8 Cytokine in Cell Supernatant After Stimulation (IFN/TNF or IL13) and Treatment (VR588, FP or CP) Conditions in ALI Cultured Epithelial Cells.
Description: Measurement of cytokine levels in cell supernatant after stimulation of isolated epithelial cells. For this study epithelial cells from severe asthma patients (n = 9) were cultured and stimulated with either IFN/TNF or IL-13 to induce inflammation. Cells are then treated with VR588 (2 concentration) or with Fluticasone Propionate (FP) or with CP690553 (CP; Tofacitinib). The concentrations of drugs are listed in the title (e.g. 10-9M).
Time Frame: 21 days
Population: 1 participant's cell did not grow
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Astma Patients
Number analyzed (Participants) | 8
pg/ml
  Non-treated Control | 2090.0 (319.7)
  Non-treated VR588 10-8M | 1835.2 (818.1)
  Non-treated VR588 10-7M | 1863.7 (310.9)
  Non-treated CP 10-7M | 1815.1 (605.1)
  Non-treated FP 10-8M | 1635.1 (530.1)
  IFN/TNF | 7000.5 (1047.4)
  IFN/TNF VR588 10-9M | 5402.1 (1427.5)
  IFN/TNF VR588 10-7M | 3996.4 (988.5)
  IFN/TNF CP 10-7M | 3050.4 (924.1)
  IFN/TNF FP 10-8M | 2558.6 (895.5)
  IL-13 | 8686.3 (2024.3)
  IL-13 VR588 10-9M | 6188.6 (734.3)
  IL-13 VR588 10-7M | 4555.2 (1467.9)
  IL-13 CP 10-7M | 4599.8 (1649.7)
  IL-13 FP 10-8M | 4639.0 (905.9)
Statistical Analysis 1: Comparison: Astma Patients; Statistical differences is determined using the Kruskal-Wallis test followed by Dunn's multiple comparison test or a Wilcoxon signed rank test as appropriate; Test type: Superiority; p = 0.0002, Wilcoxon (Mann-Whitney) — P value is the comparison between the IFN/TNF induction group versus the VR588 (10-7M) treatment group

2. Primary Outcome: Percentage of Viable Cells Compared to Baseline After Stimulation (IFN/TNF or IL13) and Treatment (VR588, FP or CP) Conditions in ALI Cultured Epithelial Cells.
Description: Measurement of cell viability after stimulation of isolated epithelial cells. For this study epithelial cells from severe asthma patients (n = 9) were cultured and stimulated with either IFN/TNF or IL-13 to induce inflammation. Cells are then treated with VR588 (2 concentration) or with Fluticasone Propionate (FP) or with CP690553 (CP; Tofacitinib). The concentrations of drugs are listed in the title (e.g. 10-9M).
Time Frame: 21 days
Population: 1 participant's cell did not grow
Measure: Mean (Standard Deviation); unit: percentage against baseline
Arm/Group | Astma Patients
Number analyzed (Participants) | 8
percentage against baseline
  Non-treated Control | 100.0 (30.1)
  Non-treated VR588 10-9M | 98.4 (23.1)
  Non-treated VR588 10-7M | 95.4 (23.2)
  Non-treated CP 10-7M | 98.4 (14.1)
  Non-treated FP 10-8M | 102.9 (27.1)
  IFN/TNF | 87.1 (10.5)
  IFN/TNF VR588 10-9M | 92.0 (15.0)
  IFN/TNF VR588 10-7M | 93.3 (14.5)
  IFN/TNF CP 10-7M | 96.6 (10.5)
  IFN/TNF FP 10-8M | 82.2 (11.2)
  IL-13 | 91.4 (12.4)
  IL-13 VR588 10-9M | 86.9 (14.2)
  IL-13 VR588 10-7M | 90.0 (10.7)
  IL-13 CP 10-7M | 89.0 (11.7)
  IL-13 FP 10-8M | 92.7 (12.4)
Statistical Analysis 1: Comparison: Astma Patients; Statistical differences is determined using the Kruskal-Wallis test followed by Dunn's multiple comparison test or Wilcoxon signed rank test as appropriate; Test type: Superiority; p = 0.3994, Wilcoxon (Mann-Whitney) — P value is the comparison between the IFN/TNF induction group versus the VR588 (10-7M) treatment group

3. Primary Outcome: Relative Fluorescence Units of STAT1 Protein Phosphorylation After Stimulation (IFN/TNF or IL13) and Treatment (VR588, FP or CP) Conditions in ALI Cultured Epithelial Cells.
Description: Measurement of activation of phospho-STAT1 member of the JAK/STAT signaltransduction pathway in cell lysates. For this study epithelial cells from severe asthma patients (n = 9) were cultured and stimulated with either IFN/TNF or IL-13 to induce inflammation. Cells are then treated with VR588 (2 concentration) or with Fluticasone Propionate (FP) or with CP690553 (CP; Tofacitinib). The concentrations of drugs are listed in the title (e.g. 10-9M).
Time Frame: 21 days
Population: 1 participant's cell did not grow
Measure: Mean (Standard Deviation); unit: Relative Fluorescence Units
Arm/Group | Astma Patients
Number analyzed (Participants) | 8
Relative Fluorescence Units
  Non-treated Control | 0.80 (0.11)
  Non-treated VR588 10-9M | 0.82 (0.13)
  Non-treated VR588 10-7M | 0.74 (0.20)
  Non-treated CP 10-7M | 0.64 (0.22)
  Non-treated FP 10-8M | 0.60 (0.28)
  IFN/TNF | 6.94 (1.75)
  IFN/TNF VR588 10-9M | 4.99 (1.82)
  IFN/TNF VR588 10-7M | 4.15 (1.55)
  IFN/TNF CP 10-7M | 1.56 (0.96)
  IFN/TNF FP 10-8M | 3.20 (1.36)
  IL-13 | 4.24 (1.72)
  IL-13 VR588 10-9M | 1.97 (1.37)
  IL-13 VR588 10-7M | 1.38 (0.71)
  IL-13 CP 10-7M | 0.89 (0.36)
  IL-13 FP 10-8M | 0.96 (0.37)
Statistical Analysis 1: Comparison: Astma Patients; Statistical difference is determined using the Kruskal-Wallis test followed by Dunn's multiple comparison test or a Wilcoxon signed rank test as appropriate; Test type: Superiority; p = 0.0104, Wilcoxon (Mann-Whitney) — P value is the comparison between the IFN/TNF induction group versus VR588 (10-7M) treatment group

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Astma Patients
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes